CLINICAL TRIAL: NCT06106893
Title: A Single-center Clinical Study Evaluating the Safety and Efficacy of CD19 Universal CAR-γδT Cells in Active Systemic Lupus Erythematosus
Brief Title: A Clinical Study of CD19 Universal CAR-γδT Cells in Active Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Qiubai Li, M.D. & Ph.D., Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230443
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; CD19 Universal CAR-γδ T Cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Participants will receive CD19 Universal CAR-γδ T Cells intravenous infusion
  Interventions: Biological: CD19 Universal CAR-γδ T Cells

INTERVENTIONS:
Biological: CD19 Universal CAR-γδ T Cells — Intravenous infusion of CD19 Universal CAR-γδ T Cells

SUMMARY:
The purpose of the study is to explore the safety and efficacy of CD19 Universal CAR-γδT cells in active severe systemic lupus erythematosus.

DETAILED DESCRIPTION:
The prognosis of patients with active systemic lupus erythematosus (SLE) remains poor, due to two major therapeutic obstacles: (1) current treatment strategies including glucocorticoids, immunosuppressive agents, biological agents, are still difficult to achieve disease control, making the disease condition of some patients continue to be active or even worse; (2) some patients are unable to wean themselves off glucocorticoid and face the risk of numerous adverse effects caused by long-term glucocorticoid dependence, such as glucocorticoid-related diabetes, femoral head necrosis, hypertension, stress ulcers, and infection, etc. Therefore, there is a strong unmet clinical need for more effective treatment for patients suffering from active SLE. Several preclinical studies have shown the efficacy of CAR-T cell treatment in SLE. The aim of this study is to investigate the safety, tolerability, preliminary efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of CD19 Universal CAR-γδT cells therapy in active SLE. Patients with active SLE will be invited to participate in the study, to receive CD19 Universal CAR-γδT cells intravenous infusion and follow-up visits of up to 2 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their guardians understand and voluntarily sign the informed consent form, and be able to complete all the documents, procedures, follow-up examinations and treatments specified in the study protocol, with good compliance;
2. Age range from 18 to 70 years old, regardless of gender;
3. Body weight ≥ 40kg;
4. Participants diagnosed with SLE according to the American College of Rheumatology (ACR) 1997 revised criteria for SLE at least 24 weeks prior to signing the informed consent form;
5. active SLE needs to meet the following criteria at screening: SELENA-SLEDAI score ≥ 6 points; PGA ≥ 1 points;
6. Have received at least 8 weeks of standardized treatment for SLE prior to screening;
7. Female participants need to have a negative pregnancy test, and participants agree to take effective contraceptive measures throughout the study.

Exclusion Criteria:

1. Known hypersensitivity to prednisone, immunosuppressive agents;
2. Diagnosis of active severe lupus nephritis within 8 weeks prior to screening, requiring medications prohibited by the research protocol for active nephritis, hemodialysis or prednisone ≥ 100 mg/d, or equivalent glucocorticoid therapy for ≥14 days;
3. Suicidal ideation within the past 6 months based on assessment by Columbia-Suicide Severity Rating Scale (C-SSRS) at screening; or any suicidal behaviors within the past 12 months or recurrent suicidal behaviors during the subject's lifetime;
4. Presence of SLE or non-SLE related central nervous system diseases or pathological changes within 8 weeks prior to screening;
5. Existence of other lupus crisis within 8 weeks prior to screening;
6. Previous or current diagnosis of non-SLE-related inflammatory arthropathy or skin diseases;
7. Previous or current diagnosis of severe vasculitis due to other diseases excluding SLE;
8. History of vital organ transplantation or hematopoietic stem cell/or bone marrow transplantation;
9. Have received plasmapheresis, hemodialysis, intravenous immunoglobulin within 14 days prior to screening;
10. Other autoimmune diseases requiring systemic therapy;
11. Active or latent tuberculosis at screening (can be enrolled if appropriately treated);
12. Any of severe laboratory abnormalities in liver function, renal function, bone marrow function, coagulation function, pulmonary function, cardiac function at screening;
13. History of severe allergy or known hypersensitivity to any of the active ingredients of the drugs, excipients, or rodent-derived products, xenoproteins included in this trial, or subjects with allergic constitution;
14. Severe heart diseases;
15. Severe hepatobiliary disease;
16. Presence of medical conditions that are obviously unstable or not effectively treated;
17. Presence of uncontrollable bacterial, fungal, viral or other infections, requiring antibiotic therapy;
18. Have received live/attenuated vaccination within 4 weeks prior to screening or plan to receive live/attenuated vaccination throughout the study;
19. Have received any commercially available Janus kinase inhibitor or Bruton tyrosine kinase inhibitor within 3 half-lives prior to screening;
20. Have received B-cell targeted therapy prior to screening;
21. Have received a biologic agent other than B-cell targeted therapy within 5 half-lives prior to screening;
22. Previous received therapies with CAR-T cells or other genetically modified T cells;
23. Have received therapeutic dose of corticosteroids within 7 days prior to leukapheresis or within 72 hours prior to infusion;
24. Subjects that have undergone major surgery within 4 weeks prior to lymph depletion or those who are scheduled to undergo major surgery during the study period, or whose surgical wounds have not fully healed prior to enrollment;
25. Subjects that have donated blood for ≥ 400mL or had significant blood loss equivalent to at least 400mL within 4 weeks prior to screening, or have received a blood transfusion within 8 weeks, or plan to donate blood during the study period;
26. History of ≥ grade 2 bleeding within 4 weeks prior to screening or need for long-term continuous anticoagulant therapy;
27. Subjects with severe mental illness;
28. Alcoholics or subjects with a history of drug abuse;
29. Female subjects who are pregnant or lactating, or intend to pursue pregnancy within 2 years after the cell infusion; male patients whose female sexual partners intend to conceive within 2 years after the cell infusion;
30. History of malignancy；
31. Patients that have contraindications to any of the study procedures or have other medical conditions that may expose them to unacceptable risk, in the judgment of the investigators and/or clinical criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Within 2 years after CD19 Universal CAR-γδT cell infusion
  Safety and tolerability will be assessed by incidence and severity of adverse events (AEs) and serious AEs (SAEs). Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) are graded by ASTCT criteria, other AEs are assessed by CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Within 2 years after CD19 Universal CAR-γδT cell infusion
  Concentration of CD19 Universal CAR-γδT cell in peripheral blood will be evaluated
Pharmacodynamics (PD) | Within 28 days after CD19 Universal CAR-γδT cell infusion
  Pharmacodynamics (PD) will be assessed by levels of cytokines (IL-2、IL-6、IL-10、IFN-γ) in peripheral blood
Proportion of subjects with SRI-4 response | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24
  SRI-4 response is defined as: 1) the Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score decrease by no less than 4 points from baseline; 2) the British Isles Lupus Assessment Group (BILAG) score with no new A domain score and no more than 1 new B domain score compared to baseline; 3) the Physician Global Assessment (PGA) score increase less than 0.3 point from baseline.
Changes in the Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  Range [0, 105]，higher score represents worse disease activity
Changes in the Physician Global Assessment (PGA) score from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  Range [0, 3]，higher score represents worse disease activity
Changes in immunological indexes from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  Serum IgA, IgG, IgE and IgM will be evaluated
Changes in level of anti-nuclear antibody (ANA) in peripheral blood from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  To evaluate SLE disease activity
Changes in level of anti-double stranded DNA (dsDNA) antibody in peripheral blood from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  To evaluate SLE disease activity
Changes in levels of complement C3 in peripheral blood from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  To evaluate SLE disease activity
Changes in levels of complement C4 in peripheral blood from baseline | Within 2 years after CD19 Universal CAR-γδT cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24)
  To evaluate SLE disease activity
Changes in levels of Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) from baseline in patients with cutaneous lupus erythematosus | Within 2 years after CD19 CAR-T cell infusion (day 14, day 28, month 3, month 6, month 9, month 12, month 18, month 24
  Range [0, 70]，higher score represents larger or more severe skin involvement

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Principal Investigator — Department of Rheumatology and Immunology, Wuhan Union Hospital
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No